CLINICAL TRIAL: NCT00833417
Title: A Pivotal Phase II, Multicenter, Single-arm, Two-cohort Trial Evaluating the Efficacy and Safety of GDC-0449 in Patients With Advanced Basal Cell Carcinoma
Brief Title: A Study Evaluating the Efficacy and Safety of Vismodegib (GDC-0449, Hedgehog Pathway Inhibitor) in Patients With Advanced Basal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHH4476g; GO01541
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2012-04-30 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Basal Cell Carcinoma
Keywords: BCC; Hedgehog Pathway Inhibitor; Hedgehog; Basal Cell Cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Neoplasms, Basal Cell | interventions — HhAntag691

ARMS (1):
- Vismodegib 150 mg (Experimental): Patients received vismodegib 150 mg orally once daily until disease progression; intolerable toxicity, most probably attributable to vismodegib; or withdrawal from the study.
  Interventions: Drug: Vismodegib 150 mg

INTERVENTIONS:
Drug: Vismodegib 150 mg — Vismodegib 150 mg was provided in hard gelatin capsules.
  Other Names: GDC-0449

SUMMARY:
This was a Phase II, single-arm, two-cohort multicenter clinical trial evaluating the efficacy and safety of vismodegib (GDC-0449) in patients with advanced basal cell carcinoma. All patients received vismodegib until evidence of progression, intolerable toxicities most probably attributable to vismodegib, or withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* For patients with metastatic basal cell carcinoma (BCC), histological confirmation of distant BCC metastasis (eg, lung, liver, lymph nodes, or bone), with metastatic disease that is Response Evaluation Criteria in Solid Tumors (RECIST) measurable using computed tomography (CT) or magnetic resonance imaging (MRI).
* For patients with locally advanced BCC, histologically confirmed disease that is considered to be inoperable.
* For patients with locally advanced BCC, radiotherapy must have been previously administered for their locally advanced BCC, unless radiotherapy is contraindicated or inappropriate. For patients whose locally advanced BCC has been irradiated, disease must have progressed after radiation.
* For women of childbearing potential, agreement to the use of two acceptable methods of contraception, including one barrier method, during the study and for 12 months after discontinuation of vismodegib (GDC-0449).
* For men with female partners of childbearing potential, agreement to use a latex condom, and to advise their female partner to use an additional method of contraception during the study and for 3 months after discontinuation of vismodegib.

Exclusion Criteria:

* Prior treatment with vismodegib or other Hedgehog pathway inhibitors.
* Pregnancy or lactation.
* Life expectancy of < 12 weeks.
* Patients with superficial multifocal BCC who may be considered unresectable due to breadth of involvement.
* Concurrent non-protocol-specified anti-tumor therapy (eg, chemotherapy, other targeted therapy, radiation therapy, or photodynamic therapy).
* Recent, current, or planned participation in an experimental drug study.
* History of other malignancies within 3 years of the first day of treatment with vismodegib in this study (Day 1), except for tumors with a negligible risk for metastasis or death, such as adequately treated squamous-cell carcinoma of the skin, ductal carcinoma in situ of the breast, or carcinoma in situ of the cervix.
* Uncontrolled medical illnesses such as infection requiring treatment with intravenous antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Hou, M.D., Study Director — Genentech, Inc.
Locations (34):
- United States (19):
  - Scottsdale, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Stanford, California
  - Aurora, Colorado
  - Ormond Beach, Florida
  - Chicago, Illinois
  - Sioux City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - New York, New York
  - Chapel Hill, North Carolina
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
- Australia (3):
  - Kogarah, New South Wales
  - Melbourne
  - Woolloongabba
- Belgium (2):
  - Brussels
  - Wilrijk
- France (4):
  - Lille
  - Nantes
  - Paris
  - Pierre-Bénite
- Germany (4):
  - Essen
  - Kiel
  - Tübingen
  - Würzburg
- United Kingdom (2):
  - London
  - Poole

REFERENCES:
- [Derived] Sekulic A, Migden MR, Basset-Seguin N, Garbe C, Gesierich A, Lao CD, Miller C, Mortier L, Murrell DF, Hamid O, Quevedo JF, Hou J, McKenna E, Dimier N, Williams S, Schadendorf D, Hauschild A; ERIVANCE BCC Investigators. Long-term safety and efficacy of vismodegib in patients with advanced basal cell carcinoma: final update of the pivotal ERIVANCE BCC study. BMC Cancer. 2017 May 16;17(1):332. doi: 10.1186/s12885-017-3286-5. PMID 28511673
- [Derived] Chang AL, Arron ST, Migden MR, Solomon JA, Yoo S, Day BM, McKenna EF, Sekulic A. Safety and efficacy of vismodegib in patients with basal cell carcinoma nevus syndrome: pooled analysis of two trials. Orphanet J Rare Dis. 2016 Sep 1;11(1):120. doi: 10.1186/s13023-016-0506-z. PMID 27581207
- [Derived] Sekulic A, Migden MR, Oro AE, Dirix L, Lewis KD, Hainsworth JD, Solomon JA, Yoo S, Arron ST, Friedlander PA, Marmur E, Rudin CM, Chang AL, Low JA, Mackey HM, Yauch RL, Graham RA, Reddy JC, Hauschild A. Efficacy and safety of vismodegib in advanced basal-cell carcinoma. N Engl J Med. 2012 Jun 7;366(23):2171-9. doi: 10.1056/NEJMoa1113713. PMID 22670903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of patients ≥ 18 years old with a histologically confirmed diagnosis of advanced basal cell carcinoma (BCC), either metastatic or locally advanced BCC. Enrollment of patients with locally advanced BCC was limited to 80 of a planned total of 100 patients. Both cohorts received the same vismodegib 150 mg treatment.
Groups:
- Metastatic BCC Cohort; Locally Advanced BCC Cohort: Patients received vismodegib 150 mg orally once daily until disease progression; intolerable toxicity, most probably attributable to vismodegib; or withdrawal from the study.
Period: Overall Study
Arm/Group | Metastatic BCC Cohort | Locally Advanced BCC Cohort
Started | 33 | 71
Completed | 0 | 0
Not Completed | 33 | 71
Not completed — Adverse Event | 5 | 16
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision to Withdraw Patient | 3 | 7
Not completed — Patient Decision to Withdraw | 4 | 23
Not completed — Sponsor Decision to Terminate Study | 1 | 2
Not completed — Disease Progression | 18 | 17
Not completed — Reason Not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metastatic BCC Cohort | Locally Advanced BCC Cohort | Total
Number analyzed (Participants) | 33 | 71 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.4) | 61.2 (16.8) | 61.4 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 32 | 41
  Male | 24 | 39 | 63

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR) Determined by the Independent Review Facility
Description: OR=complete (CR) or partial response (PR). Metastatic-CR:Disappearance of all targets. PR:≥30% decreased sum of longest diameter (SLD) of targets compared to baseline (B). Locally advanced-Response=No progressive disease (PD) and ≥30% decreased SLD from baseline (radiography [R]) or ≥30% decreased SLD from B (externally visible dimension [EVD]) or completely resolved ulceration. CR:Response with no residual BCC on tumor biopsy (otherwise response was PR). PD:Any of ≥20% increased SLD from nadir (R or EVD), new ulceration, new lesions (R or physical exam) or non-target lesion progression by R.
Time Frame: From study initiation (enrollment of first patient) through 9 months following the first treatment of the last enrolled patient (clinical cutoff date of 26 November 2010), up to 90 weeks
Population: Efficacy-evaluable population: All treated patients for whom the independent pathologist's interpretation of archival tissue or baseline biopsies was consistent with basal cell carcinoma.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Metastatic BCC Cohort | Locally Advanced BCC Cohort
Number analyzed (Participants) | 33 | 63
Percentage of participants | 30.3 [15.6 to 48.2] | 42.9 [30.5 to 56.0]

2. Secondary Outcome: Duration of Objective Response (OR) Determined by the Independent Review Facility
Description: Duration of OR was defined as the time from the initial CR or PR to the earliest documented disease progression (PD) or death. Metastatic BCC - PD: ≥ 20% increased sum of the longest diameter (SLD) of targets from nadir, or 1 or more new lesions. Locally advanced BCC - PD: any of: (1) ≥ 20% increased SLD from nadir (radiography or externally visible dimension); (2) new ulceration; (3) new lesions (radiography or physical exam); (4) progression of non-target lesions by radiography.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Metastatic BCC Cohort | Locally Advanced BCC Cohort
Number analyzed (Participants) | 10 | 27
Months | 7.6 [5.62 to NA] — The upper limit of the 95% confidence interval could not be estimated due to the small number of patients who had an objective response. | 7.6 [5.65 to 9.66]

3. Secondary Outcome: Progression-free Survival (PFS) Determined by the Independent Review Facility
Description: PFS was defined as the time from start of treatment to the earliest documented disease progression (PD) or death. Metastatic BCC - PD: ≥ 20% increased sum of the longest diameter (SLD) of targets from nadir, or 1 or more new lesions. Locally advanced BCC - PD: any of: (1) ≥ 20% increased SLD from nadir (radiography or externally visible dimension); (2) new ulceration; (3) new lesions (radiography or physical exam); (4) progression of non-target lesions by radiography.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Metastatic BCC Cohort | Locally Advanced BCC Cohort
Number analyzed (Participants) | 33 | 63
Months | 9.5 [7.36 to NA] — The upper limit of the 95% confidence interval could not be estimated due to the small number of patients with disease progression. | 9.5 [7.39 to 11.93]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the initial dose of vismodegib until death from any cause.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Metastatic BCC Cohort | Locally Advanced BCC Cohort
Number analyzed (Participants) | 33 | 63
Months | NA [NA to NA] — The data were not mature for analysis. Only 7 deaths were reported as of the 26 November 2010 data cutoff. | NA [NA to NA] — The data were not mature for analysis. Only 6 deaths were reported as of the 26 November 2010 data cutoff.

5. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36) Health Survey Scores
Description: The SF-36 Health Survey (Version 2) uses patient-reported symptoms on 8 subscales to assess health-related quality of life (HRQoL). The Physical Component Summary (PCS) score summarizes the subscales Physical Functioning, Role-Physical, Bodily Pain, and General Health. The Mental Component Summary (MCS) score summarizes the subscales Vitality, Social Functioning, Role-Emotional, and Mental Health. Each score was scaled from 0 to 100. A positive change score indicates better HRQoL.
Time Frame: Baseline, Week 12, Week 24, and at the end of the study or early termination visit, up to 90 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Metastatic and Locally Advanced BCC Cohorts: Patients received vismodegib 150 mg orally once daily until disease progression; intolerable toxicity, most probably attributable to vismodegib; or withdrawal from the study.
Arm/Group | Metastatic and Locally Advanced BCC Cohorts
Number analyzed (Participants) | 93
Units on a scale
  Change in MCS score at Week 12, n=82 | 2.20 [-0.22 to 4.62]
  Change in MCS score at Week 24, n=75 | 2.29 [0.05 to 4.53]
  Change in MCS score at end of study, n=20 | -3.80 [-10.55 to 2.96]
  Change in PCS score at Week 12, n=82 | -1.25 [-2.86 to 0.36]
  Change in PCS score at Week 24, n=75 | -1.90 [-3.75 to -0.05]
  Change in PCS score at end of study, n=20 | -2.86 [-7.39 to 1.66]

6. Secondary Outcome: Percentage of Patients With Absence of Residual Basal Cell Carcinoma (BCC) in Patients With Locally Advanced BCC
Description: In patients with locally advanced BCC, the histopathological effect of vismodegib was determined in tissue biopsies obtained at baseline and following vismodegib treatment. Reported are the percentage of patients with pathology confirmed BCC in baseline biopsy who had an absence of residual BCC post-baseline as assessed by an independent pathological review.
Time Frame: From baseline through end of the study, up to 90 weeks
Population: Efficacy-evaluable population: All treated patients for whom the independent pathologist's interpretation of archival tissue or baseline biopsies was consistent with basal cell carcinoma. Only locally advanced BCC patients with available post-baseline biopsy assessed by an independent pathologist were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Locally Advanced BCC Cohort
Number analyzed (Participants) | 51
Percentage of participants
  Total | 54.0
  Prior to Week 24 | 9.5
  At Week 24 | 42.9
  After Week 24 | 1.6

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were recorded from study initiation (enrollment of first patient) through the end of the study (09 Apr 2014).
Description: Adverse events were reported for the safety analysis population, which was defined as all enrolled patients who received any amount of study drug.
Arm/Group | Metastatic and Locally Advanced BCC Cohorts
Serious Adverse Events (participants affected / at risk) | 36/104
Other Adverse Events (participants affected / at risk) | 103/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic and Locally Advanced BCC Cohorts (N=104)
Cardiac failure (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Aphagia (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Death (General disorders) | 3
Cholestasis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 2
Meningitis viral (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Convulsion (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 4
Renal failure (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac flutter (Cardiac disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 1
Osteomyelitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic and Locally Advanced BCC Cohorts (N=104)
Anaemia (Blood and lymphatic system disorders) | 8
Nausea (Gastrointestinal disorders) | 34
Diarrhoea (Gastrointestinal disorders) | 28
Constipation (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 19
Dyspepsia (Gastrointestinal disorders) | 11
Flatulence (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 45
Asthenia (General disorders) | 10
Pain (General disorders) | 10
Nasopharyngitis (Infections and infestations) | 14
Upper respiratory tract infection (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 10
Sinusitis (Infections and infestations) | 7
Weight decreased (Investigations) | 54
Decreased appetite (Metabolism and nutrition disorders) | 29
Muscle spasms (Musculoskeletal and connective tissue disorders) | 75
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12
Dysgeusia (Nervous system disorders) | 58
Headache (Nervous system disorders) | 16
Ageusia (Nervous system disorders) | 12
Hypogeusia (Nervous system disorders) | 11
Paraesthesia (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 7
Depression (Psychiatric disorders) | 7
Anxiety (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 69
Pruritus (Skin and subcutaneous tissue disorders) | 11
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 8
Influenza like illness (General disorders) | 7
Procedural pain (Injury, poisoning and procedural complications) | 7
Actinic keratosis (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.